CLINICAL TRIAL: NCT05970666
Title: Single Arm, Prospective, Multicenter Clinical Study of TACE With Adebrelimab and Bevacizumab for Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jianbo Chen, director, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-OBU-FJ-HCC-II-012
Record Dates: First submitted 2023-07-25; First posted 2023-08-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Adebrelimab; Hepatocellular Carcinoma; Transformation; Bevacizumab; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: TACE with adebrelimab and bevacizumab

INTERVENTIONS:
Drug: TACE with adebrelimab and bevacizumab — TACE treatment once; Adebrelimab: 20mg/kg, every 3 weeks (21 days); Bevacizumab; 15mg/kg, every 3 weeks (21 days);

SUMMARY:
To evaluate the efficacy and safety of TACE combined with adebrelimab and bevacizumab transformation in unresectable hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 ~ 75, both male and female；
2. Strictly comply with the primary liver cancer diagnosis and treatment standard (2022 edition) clinical diagnosis criteria or primary hepatocellular carcinoma diagnosed by pathological histology or cytology examination, and at least one measurable lesions (according to the RECIST1.1 standard, the spiral CT scan of 10mm or short diameter of 15mm）；
3. Patients without previous systematic treatment and inoperable resection / radical ablation surgery, but who can tolerate TACE;
4. The CNLC stage is Ⅱa-Ⅲb stage;
5. The Child-Pugh grade of liver function is A grade or B grade (5-7 points);
6. The ECOG PS score is 0-1 points;
7. Expected survival period of 12 weeks;
8. If the patient has active hepatitis B virus (HBV) infection: HBV-deoxyribonucleic acid (DNA) must be <2000 IU / mL (if the study site has only copy / mL testing units, Must be <12500 copy / mL), And received at least 14 days before initiating anti-HBV treatment (according to local standard therapy, e. g. entecavir) and willing to receive antiviral treatment throughout the study; hepatitis C virus (HCV) ribonucleic acid (RNA) positive patients must receive antiviral treatment according to local standard treatment guidelines and liver function within grade CTCAE 1 elevation;
9. Main organs function are normal and meet the following criteria: (1) The blood routine examination standards should be met with: (no blood transfusion within 14 days) A. Hemoglobin (HB), 90g / L, B. White blood cell count (WBC) 3109 / L C. Absolute neutrophil count (ANC) 1.5109 / L, D. Platelet (PLT) 80109 / L;(2) Biochemical examination shall meet the following standards: A. Bilirubin (BIL) <1.5 times the upper limit of normal value (ULN); B. Glutamic gamma aminotransferase (ALT) and glutamate aminotransferase AST <5 ULN; C. Serum creatinine (Cr)≤1.5ULN；
10. Women of childbearing age must have negative pregnancy test (serum) or urine HCG within 7 days before enrollment and are willing to use appropriate contraception during treatment and 24 weeks after the last administration of test drug; for men, surgical sterilization or agree to use appropriate contraception during and 24 weeks after the last administration of trial drug;
11. The subjects volunteered to join the study and had good compliance with the follow-up.

Exclusion Criteria:

1. Pregnant or lactating women;
2. The pathology is clearly cholangiocytic carcinoma or mixed cell carcinoma;
3. Diffuse liver cancer;
4. Patients with autoimmune diseases, organ / hematopoietic stem cell transplantation or other malignant tumors (except for cured basal skin cell carcinoma and cervix carcinoma in situ);
5. Patients with consciousness disorders or unable to cooperate with the treatment, combined with patients with mental illness;
6. Patients who have participated in other clinical trials in the recent three months;
7. Previous history of other malignancies or have received targeted therapy and other PD-1 / PD-L1 inhibitor therapy;
8. Received major surgery or chemotherapy or other systemic therapy for target lesions (including not limited to radiation therapy, ablation therapy, etc.) within 1 month prior to enrollment;
9. Use of immunosuppressants or systemic hormone therapy within 14 days before enrollment to achieve immunosuppressive purposes (dose> 10mg / day prednisone or other efficacy hormones);
10. Liver function was graded as Child-Pugh C, which could not be improved by liver care treatment；
11. esophageal (gastric fundus) varices rupture and bleeding within 1 month before treatment；
12. Uncorrectable coagulopathy and severe blood abnormalities, with severe bleeding tendency. Platelet count <50109 / L and severe coagulation abnormalities against surgery (anticoagulation therapy and / or anticoagulant therapy should be stopped for more than 1 week before radiation therapy);
13. A stubborn amount of ascites, pleural fluid, malignant fluid;
14. Active infection, especially the inflammation of the biliary tract system;
15. Severe functional failure of the liver, kidney, heart, lung, brain and other major organs;
16. Previously allergic to PD-1 / PD-L1 mAb / any component of the targeted drug or other similar trials;
17. Patients with hypertension who cannot be reduced to the normal range by antihypertensive medication (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg);
18. Previous severe cardiovascular disease, including but not limited to the following diseases: myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including 450 ms in QTc men and 470 ms in women); cardiac dysfunction by NYHA, or cardiac ultrasound indicating left ventricular ejection fraction (LVEF) <50%;
19. Patients with positive urinary protein (urinary protein test of 2 + or above, or 24-hour urinary protein quantification of> 1.0g);
20. Failure to swallow tablets, malabsorption syndrome, or any condition affecting gastrointestinal absorption;
21. According to the discretion of the investigator, patients with other concomitant diseases that seriously endanger patient safety or affect the completion of the study;
22. Patients with radiotherapy, targeted therapy, and other contraindications to immunotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | Up to 2 years
  Refers to the proportion of all subjects with the best overall response (BOR) as complete remission (CR) or partial remission (PR) according to mRECIST 1.1 criteria.
Occurence of AE and SAE | Up to 2 years
  Occurence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）

SECONDARY OUTCOMES:
Radical (R0) resection rate after conversion therapy | Up to 2 years
  The cut margin had no residual cancer cells
percent conversion | Up to 2 years
  The ates of conversion to operable patients in inoperable patients
Pathological complete response rate (pCR) | Up to 2 years
  The rate of no remaining tumor cells in the excised tissue samples
Major pathological response rate (MPR) | Up to 2 years
  The ratio of the tumor cells active in the removed tissue samples is less than 10%.
Progression-free survival (PFS) | Up to 2 years
  PFS was defined as the subject's date from the date of the first dose to the date of the first documented tumor progression (as assessed by mRECIST criteria, with or without continuation of treatment) or the date of death from any cause, whichever occurred first.
Disease control rate（DCR） | Up to 2 years
  Refers to the proportion of all subjects with the best overall response (BOR) according to mRECIST criteria as complete remission (CR), partial remission (PR) and stable disease (SD).
Relapse-free survival time (RFS) | Up to 2 years
  Time from date of cure surgery to time of recurrence or death
Overall survival（OS） | Up to 2 years
  Defined as the time from the date of the first dose to the death of the subject from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Chen, Principal Investigator — The First Affiliated Hospital of Xiamen University; Feng Ye, Principal Investigator — The First Affiliated Hospital of Xiamen University; congren Wang, Study Director — Quanzhou First Hospital; Qinghe Cai, Study Director — Affiliated Hospital of Putian University; Jiafei Chen, Study Director — Putian First Hospital; Yongzhong Wang, Study Director — Sanming Second Hospital; Feng Lin, Study Director — Ningde Mindong Hospital
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China